CLINICAL TRIAL: NCT04027699
Title: Predictive Mini-bolus Fluid Responsiveness in Pediatric Septic Shock
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRECISE
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Severe Sepsis or Septic Shock in Pediatric Intensive Care Unit
Keywords: Mini-bolus challenge; fluid responsiveness; volemic expansion; pediatric septic shock; severe sepsis; microcirculation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mini-bolus (Experimental): * First injection of 2ml/kg (saline solution)
  * Second injection of 18ml/kg (saline solution)
  Interventions: Procedure: Mini-bolus

INTERVENTIONS:
Procedure: Mini-bolus — * First injection of 2ml/kg (saline solution)
  * Second injection of 18ml/kg (saline solution)

SUMMARY:
Severe sepsis and septic shock remain of particular gravity in children with a current mortality of about 20 % , despite the international prevention campaigns " survival sepsis campaign ". Septic shock associates a macrocirculatory and a microcirculatory dysfunction. The volume expansion remains the treatment of severe sepsis at the initial phase supplemented by the use of vasopressors and / or inotropes. Nevertheless , it is essential to predict the fluid responsiveness after volemic expansion because fluid overload is associated with an increased morbidity in children. In studies , the volume expansion is considered effective if it allows an increase in cardiac output of more than 15 % compared to the basal level. However, their conditions of use remain very restrictive and not applicable to most of our patients ( tidal volume ≥ 7ml / kg , PEEP sufficient , absence of cardiac arrhythmia and effective sedation ) . To date , no index can be used for all patients with invasive mechanical ventilation.

It therefore seems appropriate to develop new tests to predict the response to volume expansion in children with septic shock hospitalized in pediatric intensive care.

A recent study has validated a test to predict the response to volume expansion in adults: injection of a mini-bolus of 50 ml of saline over 10s.

The aim of the study is to evaluate the effect of mini bolus fluid to predict response to fluid expansion in pediatric septic shock.

DETAILED DESCRIPTION:
Severe sepsis and septic shock remain of particular gravity in children with a current mortality of about 20 % , despite the international prevention campaigns " survival sepsis campaign " . Septic shock associates a macrocirculatory and a microcirculatory dysfunction. The volume expansion remains the treatment of severe sepsis at the initial phase supplemented by the use of vasopressors and / or inotropes . Nevertheless , it is essential to predict the fluid responsiveness after volemic expansion because fluid overload is associated with an increased morbidity in children . In studies , the volume expansion is considered effective if it allows an increase in cardiac output of more than 15 % compared to the basal level . However , their conditions of use remain very restrictive and not applicable to most of our patients ( tidal volume > 7ml / kg , PEEP sufficient, absence of cardiac arrhythmia and effective sedation ) . To date , no index can be used for all patients with invasive mechanical ventilation .

It therefore seems appropriate to develop new tests to predict the response to volume expansion in children with septic shock hospitalized in pediatric intensive care.

A recent study has validated a test to predict the response to volume expansion in adults : injection of a mini-bolus of 50 ml of saline over 10s.

The aim of the study is to evaluate the effect of mini bolus fluid to predict response to fluid expansion in pediatric septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Baby (>28 days) or children < 15 years
2. Hospitalisation in paediatric intensive
3. Clinico-biological table compatible with severe sepsis or septic shock (likely or documented)
4. Requiring the use of invasive mechanical ventilation
5. Affiliate or beneficiary of a social security
6. Legal guardians Consent Form or Emergency Procedure

Exclusion Criteria:

1. Any serious hemodynamic clinical situation that would be delayed by inclusion in the protocol
2. Patient with shunt heart disease
3. Patient in spontaneous or non-invasive ventilation or CPAP
4. Patient with a contraindication to volemic/fluid expansion (major cardiac dysfunction, acute renal failure)
5. Patient with cardiac arrest upper 5 min
6. ECMO
7. Postcardiotomia

Ages: 28 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Cardiac output variability (ΔCO) | 5 minutes
  Cardiac output
Cardiac output variability (ΔCO) | 15 minutes
  Cardiac output : ΔCO (mL/min) = VES (ml)* heart rate and VES (cm3)= ITVA0(cm) * SA0 (cm2)

SECONDARY OUTCOMES:
Heart rate variation (ΔHR) | 15 minutes
  Heart rate usual monitoring
Systolic, diastolic and mean arterial pressure variation (ΔSAP, ΔDAP, ΔMAP) | 5 minutes
  Arterial pressure invasive or not invasive monitoring according the care of patient
Systolic, diastolic and mean arterial pressure variation (ΔSAP, ΔDAP, ΔMAP) | 15 minutes
  Arterial pressure invasive or not invasive monitoring according the care of patient
Pulse pressure variation (ΔPP) | 5 minutes
  Pulse pressure invasive or not invasive monitoring according the care of patient
Pulse pressure variation (ΔPP) | 15 minutes
  Pulse pressure invasive or not invasive monitoring according the care of patient
Systolic ejection volume variation (ΔSEV) | 5 minutes
  Systolic ejection volume is measured by transthoracic echocardiography :
  VES (ml) =ITVa0*Sa0
Systolic ejection volume variation (ΔSEV) | 15 minutes
  Systolic ejection volume is measured by transthoracic echocardiography :
  VES (ml) =ITVa0*Sa0
Velocity time-index variation (ΔVTI) | 5 minutes
  ITVA0 is measured by transthoracic echocardiography with Doppler
Velocity time-index variation (ΔVTI) | 15 minutes
  ITVA0 is measured by transthoracic echocardiography with Doppler
Microvascular Flow Index variation (ΔMFI) | 5 minutes
  Microvascular Flow Index calculated by the Microscan software (Microvision)
Microvascular Flow Index variation (ΔMFI) | 15 min
  Microvascular Flow Index calculated by the Microscan software (Microvision)
Proportion Perfused Vessels variation (ΔPPV) | 5 minutes
  Proportion Perfused Vessels calculated by the Microscan software (Microvision)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Dupic, MD, Study Chair — APHP
Locations (1):
- Hôpital Necker Enfants-Malades, Paris, France